CLINICAL TRIAL: NCT05535062
Title: A Prospective, Randomized, Single Blind, Crossover Study to Evaluate Treatment Effects Associated With the NeuroStar New Treatment Feature
Brief Title: Study to Evaluate Treatment Effects Associated With the NeuroStar SoftStart Treatment Feature
Acronym: Comfort Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 44-03054-000
Record Dates: First submitted 2022-09-01; First posted 2022-09-10 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder
Keywords: TMS; Major Depressive Disorder; NeuroStar TMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will be switched between different treatment arms and asked to complete questionnaires.
Who Masked: Participant
Masking Description: The study will be randomized to avoid any bias in treatment arm assignment. Subjects will be blinded to the actual treatment arm throughout the study to allow patient to provide an honest assessment of the treatment they are receiving daily. Subjects will not be informed of the treatment at the end of their study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dash protocol ramp first (Active Comparator): Patients will be randomized after consent to receive a standard Dash protocol ramp. After the ramping phase, participants will receive both active conditions in the order: modified protocol, dash, modified protocol, dash. Protocols will be delivered 24 hours apart.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Modified Dash protocol ramp first (Active Comparator): Patients will be randomized after consent to receive a modified Dash protocol ramp. After the ramping phase, participants will receive both active conditions in the order: dash, modified protocol, dash, modified protocol. Protocols will be delivered 24 hours apart.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — the administration of a series of magnetic stimuli to the brain for the purpose of altering brain function

SUMMARY:
The purpose of this study is to evaluate the comfort of the NeuroStar® Advanced Therapy System regular prescribed TMS protocol versus a New Feature.

DETAILED DESCRIPTION:
This is a 2 week study to evaluate the New Feature an exclusive feature available on the NeuroStar® Advanced Therapy System. This feature introduces a series of stepped pulses within each pulse train ramping up the pulse magnitude to the prescribed treatment level. Patients will be randomized after consent to receive either the standard Dash protocol or the modified Dash protocol with the New feature enabled. The subjects will be switched between treatment protocols and asked to complete comfort, and depression questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 1. 22-70 years.
* 2. Subject qualifies to receive TMS Therapy with the NeuroStar Advanced Therapy System to treat Major Depressive Disorder (MDD) per current FDA-cleared treatment guidelines as evaluated by the treating physician.

  3. Subject has MDD diagnosis according to applicable DSM-IV, DSM-IV-TR, DSM-V, ICD-9, or ICD-10 criteria.

  4. Subject failed to respond to at least one prior anti-depressant medication. 5. Subject consented to receive TMS Therapy to treat MDD with his or her physician independent of potential participation in this clinical study.

  6. Subject must agree not to take analgesic pain medication(s) within 8 hours prior to TMS therapy sessions.

  7. Subject provides written consent to take part in the study.

Exclusion Criteria:

* 1. Subject satisfies any one or more of the contraindications for TMS Therapy per current treatment guidelines as determined by the PI.

  2. Physician intends to treat the subject with an off-label TMS Therapy or indication.

  3. Family history of seizures or epilepsy. 4. Subject has received prior TMS. 5. Subject is currently taking analgesic medication or substances which may affect their perception or sensation of pain.

  6. Known or suspected pregnancy.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve A Erickson, BS, Study Director — Neuronetics
Locations (1):
- TMS of South Tampa, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified DASH First: Participants started with modified dash protocols first.
- DASH Treatment First: Participants started with DASH treatment first
Period: Ramp up Phase (5 Days)
Arm/Group | Modified DASH First | DASH Treatment First
Started | 17 | 23
Completed | 17 | 23
Not Completed | 0 | 0
Period: Treatment Phase (4 Days)
Arm/Group | Modified DASH First | DASH Treatment First
Started | 17 | 23
Completed | 17 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Patients will be randomized after consent to receive modified Dash protocol with the New feature enabled
  repetitive Transcranial Magnetic Stimulation: the administration of a series of magnetic stimuli to the brain for the purpose of altering brain function
Arm/Group | All Subjects
Number analyzed (Participants) | 40
Age, Customized [Mean (Full Range); unit: years]
  Mean Age | 42 [22 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 6
Primary diagnosis [Count of Participants; unit: Participants] — Primary Diagnosis of F33.2 Major Depressive Disorder
  Participants | 40

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Comfort of TMS Treatment
Description: The average Visual Analog Scale scores for the two conditions Dash protocol and modified DASH.
  VAS - Visual Analog Scale range is 0-100 (0- no pain/discomfort; 100- extreme discomfort/worse pain)
Time Frame: 10 days
Population: VAS scores were collected for both standard and modified dash conditions for each participant. An average VAS score for each condition was calculated for each participant.
Measure: Mean (Standard Deviation); unit: VAS score on a scale
Groups:
- Modified DASH: All participants receiving Modified DASH condition
- DASH: All participants receiving DASH condition
Arm/Group | Modified DASH | DASH
Number analyzed (Participants) | 40 | 40
VAS score on a scale | 29.9 (18.4) | 29.3 (18.0)

2. Secondary Outcome: Time to Reach Prescribed Treatment Intensity
Description: Th average time to reach the prescribed treatment intensity. Once TMS therapy begins, adjustments to the stimulation intensity can begin immediately, as needed, according to subject tolerance. The TMS treater will assess if the subject can tolerate escalating the treatment MT by 10% at different time points. At each interval and the end of treatment, the treater will record the current intensity (%MT) achieved. The goal will be to reach and sustain the target intensity established by the treating physician (120%MT).
Time Frame: 5 days
Population: Average time in number of days to reach maximum treatment intensity (120% MT). During the ramp-up phase, this could take 1-5 days in both arm.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Dash Protocol Ramp: Patients will be randomized after consent to receive standard Dash protocol ramp
- Modified Dash Protocol Ramp: Patients will be randomized after consent to receive modified Dash protocol ramp using the new enabled feature
Arm/Group | Dash Protocol Ramp | Modified Dash Protocol Ramp
Number analyzed (Participants) | 23 | 17
days | 1.78 (1.28) | 1.9 (1.05)

ADVERSE EVENTS:
Time Frame: up to 9 days for each subject. 1st day of treatment to last day of treatment
Description: Standard adverse event definition
Groups:
- Dash Protocol: Patients will be randomized after consent to receive standard Dash protocol
  repetitive Transcranial Magnetic Stimulation: the administration of a series of magnetic stimuli to the brain for the purpose of altering brain function
- Modified Dash Protocol With the New Feature Enabled: Patients will be randomized after consent to receive modified Dash protocol with the New feature enabled
  repetitive Transcranial Magnetic Stimulation: the administration of a series of magnetic stimuli to the brain for the purpose of altering brain function
Arm/Group | Dash Protocol | Modified Dash Protocol With the New Feature Enabled
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 4/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dash Protocol (N=40) | Modified Dash Protocol With the New Feature Enabled (N=40)
Eye Discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand Movement (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (4) — During TMS, subject reported involuntary hand movement that was corrected by coil adjustment.
Discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT05535062/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT05535062/SAP_001.pdf